CLINICAL TRIAL: NCT05078996
Title: Patient-Centred Care and Treatment-related Quality of Life With Infertility
Brief Title: Treatment-related Quality of Life and Patient-Centred Care With Infertility
Status: Completed | Type: Observational
Sponsor: Elif Balkan (Other)
Responsible Party: Sponsor-Investigator, Elif Balkan, Master of Science, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: Istanbul UC
Record Dates: First submitted 2021-06-19; First posted 2021-10-15 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Patient Centred Care; Compliance, Treatment; Infertility, Female; Quality of Life
Keywords: patient centred care; FertiQol; infertility; quality of life; nursing
MeSH Terms: conditions — Patient Compliance; Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted in a cross-sectional descriptive type with 160 infertile women who were treated in the IVF Clinic of a university hospital between July - October 2020 in order to evaluate the effect of patient-centered care approach in infertility on treatment-related quality of life. The data of the study were collected face to face through the "Introductory Information Form" "Patient Centered Care Form for Infertile Women" and "FertiQol Treatment Module".

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with infertility
* Has no commnunication problems

Exclusion Criteria:

* Communication problems (e.g language)
* Diagnosed by diseases with reproductive problems but not infertility

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who diagnosed with infertility
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment-related quality of life | from obtaining ethical permission to reaching sampling (approximately 6 months)
  FertiQol Treatment Module was used to evaluate treatment-related quality of life. This module is a sub-module within FertiQol Scale which developed by Boivin et al. (2011). Module has 10 questions about treatments physical and emotional effects. Module has two subdimensions called "Environment" and "Tolerability" and each subdimensions and total scale score can between 0-100 points.

SECONDARY OUTCOMES:
Patient Centred Care | from obtaining ethical permission to reaching sampling (approximately 6 months)
  Patient Centred Care Questionnaire Form for Infertile Women was used to evaluate patient centred care approach. This questionnaire was prepared by researchers according to literature (IOM, 2001; Picker, 2001).There is no scoring for this tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Balkan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No